CLINICAL TRIAL: NCT02847728
Title: Pattern of Use and Safety/Effectiveness of Nivolumab in Routine Oncology Practice
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-234
Record Dates: First submitted 2016-06-28; First posted 2016-07-28 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Melanoma; Lung Cancer
MeSH Terms: conditions — Melanoma; Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single Arm Design: The study encompasses a single arm design with 417 adults treated with nivolumab for histologically or cytologically confirmed melanoma and 772 adults treated with nivolumab for histologically or cytologically confirmed lung cancer.

SUMMARY:
This is an observational, multicenter study in participants treated with nivolumab for the approved indications of melanoma and Lung cancer in Australia, the EU, Switzerland, the United Kingdom (UK), and the United States (US). The targeted countries in the EU for study participation include Austria, Belgium, Czech Republic, France, Germany, Hungary, Italy, Poland, and Spain. Study objectives are to assess the safety experience, survival, adverse event management, and outcomes of adverse events associated with nivolumab in routine oncology care facilities.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Histologically or cytologically confirmed diagnosis of melanoma (including uveal melanoma) or lung cancer
* Treatment with commercial nivolumab for the first time, alone or in combination with ipilimumab, for the approved indications of nivolumab within 14 days before informed consent for this study OR in the case where treatment has not yet been initiated, documentation that the treatment strategy is determined before an informed consent to study participation, and treatment is initiated within 28 days after informed consent

Exclusion Criteria:

* Prior participation in a clinical trial within the past 4 weeks
* Previously treated with anti-PD-1, anti-PD-L1, or anti-PD-L2 antibodies
* Previously treated with anti-CTLA-4 for lung cancer
* Current or pending participation in a clinical trial
* Current or pending systemic treatment for cancer other than melanoma and lung cancer
* Inability to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of 417 adults treated with nivolumab for histologically or cytologically confirmed melanoma and 772 adults treated with nivolumab for histologically or cytologically confirmed lung cancer in accordance with the approved indications in Australia, the EU, Switzerland, the UK, and the US. The targeted countries in the EU for participant enrollment include Austria, Belgium, Czech Republic, France, Germany, Hungary, Italy, Poland, and Spain. Participants who begin treatment with nivolumab for the first time will be enrolled in accordance with the approved indications and whose treatment strategy was determined independently from consideration of study participation. Treatment will be determined at the treating physician's discretion and with the participant's consent.
Sampling Method: Probability Sample
Enrollment: 1189 (Actual)
Dates: Start 2016-07-28 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence rate of and severity of immune-related pneumonitis - Melanoma | up to nine years
Incidence rate of and severity of immune-related colitis- Melanoma | up to nine years
Incidence rate of and severity of immune-related hepatitis - Melanoma | up to nine years
Incidence rate of and severity of immune-related nephritis/renal dysfunction - Melanoma | up to nine years
Incidence rate of and severity of immune-related endocrinopathies - Melanoma | up to nine years
Incidence rate of and severity of immune-related rash (including toxic epidermal necrolysis) - Melanoma | up to nine years
Incidence rate of and severity of other immune-related adverse events (eg, uveitis, pancreatitis, demyelination, Guillain-Barre Syndrome, myasthenic syndrome, and encephalitis) - Melanoma | up to nine years
Incidence rate of and severity of severe infusion reactions- Melanoma | up to nine years
Incidence rate of and severity of immune-related pneumonitis - Lung Cancer | up to nine years
Incidence rate of and severity of immune-related colitis - Lung Cancer | up to nine years
Incidence rate of and severity of immune-related hepatitis - Lung Cancer | up to nine years
Incidence rate of and severity of immune-related nephritis/renal dysfunction - Lung Cancer | up to nine years
Incidence rate of and severity of immune-related endocrinopathies - Lung Cancer | up to nine years
Incidence rate of and severity of other immune related adverse events (eg, uveitis, pancreatitis, demyelination, Guillain-Barre Syndrome, myasthenic syndrome, and encephalitis) - Lung Cancer | up to nine years
Incidence rate of and severity of severe infusion reactions - Lung Cancer | up to nine years
Incidence rate of and severity of immune-related rash (including toxic epidermal necrolysis), - Lung Cancer | up to nine years

SECONDARY OUTCOMES:
Adverse Events | Up to nine years
  Other nivolumab treatment-related AEs
Management of Immune-related AEs: | Up to nine years
Outcomes of Immune-related AEs: | Up to nine years
Overall Survival: | Up to nine years
  1-, 2-, 3-, 4-, and 5-year overall and median survival
Nivolumab treatment pattern | Up to nine years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (94):
- United States (12):
  - Local Institution - 1909, Palm Springs, California
  - Local Institution - 1912, Jacksonville, Florida
  - Local Institution - 1907, Lake City, Florida
  - Local Institution - 1901, Park Ridge, Illinois
  - Local Institution - 1910, Alexandria, Louisiana
  - Local Institution - 1906, Tupelo, Mississippi
  - Local Institution - 1908, Kansas City, Missouri
  - Local Institution - 1911, Morristown, New Jersey
  - Local Institution - 1902, Bethlehem, Pennsylvania
  - Local Institution - 1913, Hilton Head Island, South Carolina
  - Local Institution - 1915, El Paso, Texas
  - Local Institution - 1905, Fort Sam Houston, Texas
- Australia (5):
  - Local Institution - 1001, Lismore, New South Wales
  - Local Institution - 1002, Wagga Wagga, New South Wales
  - Local Institution - 1006, Franskton, Victoria
  - Local Institution - 1003, Wodonga, Victoria
  - Local Institution - 1005, Subiaco, Western Australia
- Austria (3):
  - Local Institution - 1103, Innsbruck
  - Local Institution - 1102, Klagenfurt
  - Local Institution - 1101, Krems
- Belgium (3):
  - Local Institution - 1202, Brasschaat, Antwerpen
  - Local Institution - 1203, Kortrijk
  - Local Institution - 1201, Namur
- Local Institution - 2002, Olomouc, Czechia
- France (6):
  - Local Institution - 1307, Lyon
  - Local Institution - 1301, Metz-Tessy
  - Local Institution - 1305, Nancy
  - Local Institution - 1304, Saint Jean Priest En Jarez
  - Local Institution - 1303, Toulouse
  - Local Institution - 1302, Vandœuvre-lès-Nancy
- Germany (36):
  - Local Institution - 1429, Heidelberg, Baden-Wurttemberg
  - Local Institution - 1430, Greifswald, Mecklenburg-Vorpommern
  - Local Institution - 1434, Koblenz, Rheinland Pfa
  - Local Institution - 1401, Quedlinburg, Saxony-Anhalt
  - Local Institution - 1410, Lübeck, Schleswig-Holstein
  - Local Institution - 1403, Augsburg
  - Local Institution - 1423, Ballenstedt
  - Local Institution - 1427, Berlin
  - Local Institution - 1411, Bochum
  - Local Institution - 1436, Bonn
  - Local Institution - 1413, Bremerhaven
  - Local Institution - 1407, Buxtehude
  - Local Institution - 1419, Cologne
  - Local Institution - 1417, Erfurt
  - Local Institution - 1416, Gera
  - Local Institution - 1428, Giessen
  - Local Institution - 1422, Hamburg
  - Local Institution - 1424, Hamburg
  - Local Institution - 1408, Jena
  - Local Institution - 1406, Kassel
  - Local Institution - 1425, Leipzig
  - Local Institution - 1432, Ludwigshafen
  - Local Institution - 1433, Mainz
  - Local Institution - 1426, Mainz
  - Local Institution - 1405, Minden
  - Local Institution - 1431, München
  - Local Institution - 1409, München
  - Local Institution - 1420, Münster
  - Local Institution - 1418, Recklinghausen
  - Local Institution - 1402, Regensburg
  - Local Institution - 1415, Rostock
  - Local Institution - 1421, Rostock
  - Local Institution - 1435, Saarbrücken
  - Local Institution - 1414, Schwerin
  - Local Institution - 1404, Traunstein
  - Local Institution - 1412, Ulm
- Hungary (5):
  - Local Institution - 2101, Gyöngyössolymos, Heves County
  - Local Institution - 2107, Budapest
  - Local Institution - 2102, Debrecen
  - Local Institution - 2106, Farkasgyepű
  - Local Institution - 2103, Törökbálint
- Italy (6):
  - Local Institution - 1501, Bari
  - Local Institution - 1506, Lecce
  - Local Institution - 1505, Lucca
  - Local Institution - 1503, Napoli
  - Local Institution - 1502, Ravenna
  - Local Institution - 1504, Udine
- Poland (3):
  - Local Institution - 2201, Opole, Opole Voivodeship
  - Local Institution - 2202, Gdansk
  - Local Institution - 2203, Olsztyn
- Local Institution - 1904, Bayamón, Puerto Rico
- Spain (7):
  - Local Institution - 1606, Ávila
  - Local Institution - 1605, Cáceres
  - Local Institution - 1602, Jaén
  - Local Institution - 1601, Madrid
  - Local Institution - 1604, Salamanca
  - Local Institution - 1607, Santander
  - Local Institution - 1603, Toledo
- Switzerland (2):
  - Local Institution - 1703, Baden, Canton of Aargau
  - Local Institution - 1702, Locarno
- United Kingdom (4):
  - Local Institution - 1803, Aberdeen, Aberdeenshire
  - Local Institution - 1802, Truro, Cornwall
  - Local Institution - 1804, Glasgow, Strathclyde
  - Local Institution - 1801, Bristol

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome